CLINICAL TRIAL: NCT01753284
Title: Patients and Carers Experiences With First Episode Psychosis and Pathway to Care in Nordland: A Qualitative Study
Brief Title: First Episode Psychosis and Pathway to Care in Nordland
Status: Completed | Type: Observational
Sponsor: Nordlandssykehuset HF (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/1650(REK)
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Last update posted 2019-05-13 (Actual); Status verified 2018-04

CONDITIONS: First Episode Psychosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
First episode psychosis patients often experiences treatment delay. This reduces their prospects for recovery and makes unnecessary burdens for them and their carers. A better understanding of help seeking intentions is required, and has not been explored in a county like Nordland, Norway, with long distances and challenging access to health services. The purpose of this study is to explore the process of help seeking, including how patients and their careers discover and understand the psychotic symptoms. Research exploring the impact on families mainly focuses on parents' experiences, and there are less studies focusing on experiences and needs of siblings. This study will therefore explore siblings' experiences separate from their parents. Methods will be qualitative interviews with patients, their carers and siblings. Analysis will be influenced by Grounded theory.

ELIGIBILITY:
Inclusion Criteria:

* age 16-35,
* understand and speak Norwegian
* able to give consent
* no learning disabilities

Exclusion Criteria:

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients experiencing first and multiple episode psychosis carers siblings
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2018-10 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Patient experience | up to 100 weeks
Carers experiences | up to 100 weeks
Siblings experiences | up to 100 weeks
Pathway to care | up to 100 weeks